CLINICAL TRIAL: NCT01139645
Title: The Effect of Proton Pump Inhibitors on Calcium and Bone Metabolism: A Prospective Single-Blind Matched Controlled Study
Brief Title: The Effect of Proton Pump Inhibitors on Calcium and Bone Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Ala'a Sharara, Professor, American University of Beirut Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: IM.AS1.24
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Calcium Metabolism Disorders
Keywords: Calcium; bone; metabolism; Proton Pump Inhibitors; Rabeprazole; Esomeprazole; Lanzoprazole; Vitamin D; bone and bones
MeSH Terms: conditions — Calcium Metabolism Disorders | interventions — Rabeprazole; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proton Pump Inhibitors (Experimental): patients were started on Proton Pump inhibitors for 3 months (the whole duration of the study)
  Interventions: Drug: Rabeprazole or Esomeprazole or Lanzoprazole
- No Proton Pump Inhibitors (No Intervention): patients are not taking any Proton Pump Inhibitor, and they are matched by age to patients in the experimental group.

INTERVENTIONS:
Drug: Rabeprazole or Esomeprazole or Lanzoprazole — 1/3 of the patients are taking Pariet (Rabeprazole) 20 mg once daily 1/3 of the patients are taking Nexium (Esomeprazole) 40 mg once daily 1/3 of the patients are taking Lanzor (Lanzoprazole) 30 mg once daily
  Arms: Proton Pump Inhibitors

SUMMARY:
This prospective, single-blind, matched controlled study aims to evaluate the effect of proton pump inhibitors on biochemical markers of calcium and bone metabolism in an effort to establish additional biological plausibility for the apparent association between proton pump inhibitors (PPIs) and osteoporosis-related fractures.

Young males (age 18-45 years), who are either healthy volunteers, or who complain of daily or frequent heartburn but are otherwise healthy, will be recruited and enrolled in the study. Patients with heartburn will be assigned to the intervention group and will be assigned to take a PPI for three months. Healthy volunteers will be matched by age to patients in the intervention group and will act as the control group. 70 patients will be enrolled in total. Blood studies for all subjects will be taken at 0, 1 and 3 months to test for various biochemical markers of calcium and bone metabolism, which act as surrogate markers of calcium absorption and bone remodeling.

Levels of biochemical markers in the two groups will be compared using two-way analysis of variance (ANOVA). Changes in biochemical parameters within a group will be assessed using repeated measures ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-50 years
* Healthy (or healthy with heartburn only)

Exclusion Criteria:

* Female gender
* Previous allergy to PPI
* Regular beach seekers (more than once a week)
* Intestinal disease
* Recent fracture (within the past six months)
* Kidney stones
* Intake of the following medications:

  * Vitamin D or calcium supplements
  * PPIs or H2 receptor antagonists within the past year
  * One-Alpha
  * Anticonvulsants
  * Glucocorticoids

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
changes in Parathyroid hormone levels | baseline and 3 months
  PTH levels at 3 months minus at baseline

SECONDARY OUTCOMES:
changes in 25-OH-Vitamin D blood levels | baseline and 3 months
  25-OH-Vitamin D blood levels at 3 months minus baseline
changes in osteocalcin levels in blood | baseline and 3 months
  osteocalcin levels at 3 months minus at baseline
changes in crosslaps levels in blood | baseline and 3 months
  crosslaps levels in blood at 3 months minus at baseline
changes in serum ionized calcium levels | baseline and 3 months
  serum ionized calcium levels at 3 months minus at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ala' I. Sharara, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut - Medical Center, Beirut, Lebanon

REFERENCES:
- [Derived] Sharara AI, El-Halabi MM, Ghaith OA, Habib RH, Mansour NM, Malli A, El Hajj-Fuleihan G. Proton pump inhibitors have no measurable effect on calcium and bone metabolism in healthy young males: a prospective matched controlled study. Metabolism. 2013 Apr;62(4):518-26. doi: 10.1016/j.metabol.2012.09.011. Epub 2012 Oct 24. PMID 23102518